CLINICAL TRIAL: NCT05066464
Title: Fluid Resuscitation for Suspected Sepsis in Paediatric Emergency Departments (FRESSPED): a French Multicenter Prospective Observational Study
Brief Title: Fluid Resuscitation for Suspected Sepsis in Paediatric Emergency Departments
Acronym: FRESSPED
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHPHLJ
Record Dates: First submitted 2021-09-22; First posted 2021-10-04 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2021-09

CONDITIONS: Septic Shock
Keywords: Paediatric sepsis, SSC-2020, fluid bolus therapy
MeSH Terms: conditions — Shock, Septic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Fluid Resuscitation — Fluid Resuscitation for Suspected Sepsis in Paediatric Emergency Departments

SUMMARY:
With 25.2 million children affected and 3.4 million deaths in 2017, paediatric sepsis is the leading cause of under-five mortality worldwide and has recently been described as "significant global health threat" by the World Health Organization. In addition to early antibiotics, fluid bolus therapy (FBT) is one of the cornerstones of management, due to the theoretical improvement of cardiac output, oxygen delivery and organ perfusion. In the absence of a consensual and operational definition to date, the latest international guidelines of the Surviving Sepsis Campaign 2020 (SSC-2020), refers to children (≥ 37 weeks gestation at birth to 18 years old) with severe infection leading to cardiovascular (i.e., "septic shock") or non-cardiovascular organ dysfunction (i.e., "other sepsis-associated organ dysfunction" or former "severe sepsis"). The SSC-2020 specifies the modalities for paediatric sepsis management, particularly concerning FBT, with, for example, the preferential use of balanced crystalloids, and a target volume of 40-60ml/kg at one hour of recognition using boluses of 10-20ml/kg in children who have access to a paediatric intensive care unit (PICU) in their health system. Further, it is now well established that compliance with international guidelines is associated with improved outcomes in paediatric sepsis. Despite the importance of awareness and implementation of the SSC-2020, there are, to our knowledge, no studies evaluating its application in children. We prospectively conducted the Fluid Resuscitation for Suspected Sepsis in Paediatric Emergency Departments (FRESSPED) study in 25 hospitals over five weeks between November 2021 and March 2022, whose principal objective was to assess doctors adherence to the SSC-2020 guidelines when performing FBT in infants and children with suspected sepsis in French paediatric emergency departments.

DETAILED DESCRIPTION:
FRESSPED study was conducted over 5 weeks, the last week of each month, between November 2021 and March 2022 (11/29 - 12/05 ; 12/27 - 01/02 ; 01/24 - 30/01 ; 02/21 - 02/27 ; 03/21 - 03/27). Patients were followed up one month after inclusion, extending the study period until midnight on 28 April 2022.

FRESSPED study was conducted in three stages :

1. Evaluation of usual fluid bolus therapy practice in infants and children with suspected sepsis in French paediatric emergency departments, through the prospectively anonymous completion of a paper case report form (CRF) designed to be completed in less than 5 minutes, within 72 hours of inclusion, by each doctor in one of the participating centers caring for an eligible patient
2. Questioning of participating doctors at the end of the 5-week prospective data collection period, to explore the underlying reasons of doctors non-adherence to the SSC-2020 guidelines. It will take the form of a short, anonymized and blinded of centers outcomes, online survey to assess attitudes and knowledge, without inter-center or inter-individual comparisons (except for doctors seniority)
3. Description of characteristics and outcomes of included patients, by consultation, up to 1 month after inclusion, of data collected in routine care (patient chart) by the lead researcher (Julian San GEROTEO).

In addition to the above criteria, the suspicion of sepsis was confirmed retrospectively in doubtful or non-documented cases or those without microbiological documentation, using an adjudication committee composed of two medical experts particularly important in the absence of a ""gold standard"" definition of paediatric sepsis to date.

ELIGIBILITY:
Inclusion Criteria:

* Newborns (discharged from the maternity ward after full-term birth or over 39 SA corrected age) and children (under 18 years of age) admitted to the UAS of a participating center during the study period.
* Suspected sepsis according to the American Academy of Pediatrics criteria (at least 3 of the 8 criteria or 2 if high-risk patient* among dysthermia, hypotension, tachycardia, polypnea, abnormalities in CRT, pulse rate, skin and neurological examination) and blood cultures or anti-infectives prescribed within 72 hours.

  * Cancer, severe encephalopathy (non walking, non communicating), central line and immunosuppression (marrow or organ transplantation, asplenia including sickle cell disease, neutropenia, constitutional immune deficiency&) immunosuppressive or immunomodulatory treatment including corticoids within 6 months)
* Having received at least one RV (at least 5ml/kg of crystalloids or colloids in less than 60 min or of 60 min or identified as such in the patient's medical record)

Exclusion Criteria:

* Parent (or legal guardian) objection to data collection.

Ages: 1 Day to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Infants and children from paediatric emergency departments
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2021-11-29 (Actual); Primary Completion 2022-03-27 (Actual); Study Completion 2022-04-28 (Actual)

PRIMARY OUTCOMES:
Adherence to the SSC-2020 guidelines of fluid bolus therapy according to the following indicator | 1 day
  Volume of 10ml/kg to 20ml/kg for each bolus (yes/no)
Adherence to the SSC-2020 guidelines of fluid bolus therapy according to the following indicator | 1 day
  Total volume of 40-60 ml/kg of during the first hour of sepsis recognition (yes/no)
Adherence to the SSC-2020 guidelines of fluid bolus therapy according to the following indicator | 1 day
  Use of balanced crystalloids (yes/no)

CONTACTS AND LOCATIONS:
Overall Officials: Stephane DAUGER, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Robert Debre Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] San Geroteo J, Levy M, Bailhache M, De Jorna C, Privat E, Gasmi O, Fuentes-Lopez M, Laoudi Y, Mazeghrane M, Malterre A, Bories P, Abdel Aal K, Arjoca I, Gaschignard J, Tanchaleune D, Minodier P, Audren F, Mazetier T, Quagliaro P, Raimond F, Sieng S, Robert B, Wohrer D, De Suremain N, Dauger S. Assessment of adherence to the 2020 Surviving Sepsis Campaign guidelines for fluid resuscitation in children with suspected septic shock in paediatric emergency departments: a prospective multicentre study. Arch Dis Child. 2024 Jul 18;109(8):636-641. doi: 10.1136/archdischild-2023-325837. PMID 38499323